CLINICAL TRIAL: NCT01995565
Title: Impact of Systemic Hemodynamic Changes on Cerebral Perfusion and Oxygenation
Brief Title: Regional Cerebral Hemodynamics Related to Global Hemodynamics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dorothea Closhen, MD, Johannes Gutenberg University Mainz
Other Study IDs: CLS_002; 837.437.11(7979) (Other: Ethics Commitee of Rhineland Palatinate)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2011-07

CONDITIONS: Critically Ill Patients

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PLR
  Other Names: To test fluid responsiveness passive leg raising is performed

SUMMARY:
This prospective investigation studies changes in regional cerebral hemodynamics and oxygenation as a function of cardiac output and blood pressure in intensive care patients.

DETAILED DESCRIPTION:
Cerebral blood flow velocity (as an index of regional perfusion), dynamic cerebral autoregulation and regional cerebral oxygen saturation should be monitored if disturbances of cerebral perfusion and oxygenation have to be suspected. Noninvasive monitoring techniques are established. When detected early, disturbed perfusion and oxygenation may be treated promptly and permanent damage of brain tissue can be avoided.

In critically ill patients, hemodynamic changes occur due to the disease itself but also as a function of diagnostic and therapeutic procedures. Systemic hemodynamic changes can be monitored using PiCCO® system (pulse contour cardiac output, Pulsion Medical Systems, Munich, Germany) that combines transpulmonal thermodilution and pulse contour analysis. PiCCO® continuously monitors cardiac output (CO), as well as static parameters like global enddiastolic blood volume index (GEDVI), and dynamic parameters as difference in pulse pressure (dPP) and stroke volume variation (SVV), respectively. CC Nexfin® (BMeye, Amsterdam, The Netherlands) is a noninvasive hemodynamic monitor.

This study investigates the effects of changes in cardiac output on cerebral blood flow velocity and regional cerebral oxygen saturation in intensive care patients that underwent major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* critically ill
* mechanically ventilated
* needing advanced hemodynamic monitoring (PiCCO)

Exclusion Criteria:

* <18years
* > 80years
* rhythm other than sinus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
cerebral blood flow velocity | 1 hour

SECONDARY OUTCOMES:
Cerebral oxygen saturation | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg University Mainz, Mainz, Germany